CLINICAL TRIAL: NCT05114005
Title: Dance-Based Avenues to Advance Nonpharmacologic Treatment of Chemotherapy Effects (DAANCE)
Brief Title: Tango for Neuropathy Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lise Worthen-Chaudhari, Research Scientist, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015C0090; NCI-2018-00310 (Registry Identifier: CTRP); R21AG068831 (NIH); OSU-15047 (Other: Ohio State University Comprehensive Cancer Center)
Record Dates: First submitted 2021-09-20; First posted 2021-11-09 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer, Breast; Neuropathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tango (Experimental): The intervention will consist of 16 Argentine Tango (Tango) sessions, adapted for neurorehabilitation per Hackney and Earhart (2010). Delivered over 8 weeks at a frequency of 2x per week and duration of 1 hour per session, this program teaches the basics steps of partnered Tango dance.
  Interventions: Behavioral: Rhythmic Auditory Stimulation
- Home Exercise (HEX) (Active Comparator): The control group will consist of an evidence-based, structured home exercise program (HEX) based on the 8 week intervention described by Zimmer et al (2018) and recommended by physical therapists specializing in BC within our organization. This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hour training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
  Interventions: Behavioral: Evidence-Based Exercise

INTERVENTIONS:
Behavioral: Rhythmic Auditory Stimulation — Rhythmically-entrained sensorimotor activity.
  Arms: Tango
Behavioral: Evidence-Based Exercise — This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hour training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
  Arms: Home Exercise (HEX)

SUMMARY:
Group dance classes have been found to improve markers of quality of life and physical health (i.e., balance) among some populations engaged in rehabilitation, such as the elderly and individuals with Parkinson Disease. However, such interventions have yet to be studied among cancer survivors despite the relevance of quality of life and physical health within cancer survivorship. Group dance classes are a promising avenue in that they deliver activity-based medicine in a social context, thus potentially improving physical as well as psychosocial aspects of health. To further this avenue of inquiry, we propose to study the effect of dance-based interventions for cancer survivors.

DETAILED DESCRIPTION:
Participants will be randomized (1:1) to one of two activity intervention arms: Argentine Tango dance or home exercise. Information about neuropathy symptoms, motion, falls incidence, and participant feedback about the interventions will be collected.

Aim1: To evaluate change in postural control over 16 sessions of Tango (exp) vs HEX (control) (n=26 per group) as primary endpoint. As secondary measures, to assess: balance function (i.e., TUG) and patient-reported outcomes (PROs) (i.e., symptoms, pain, fatigue, mood, quality of life) monthly including 1 month post-intervention completion; postural control and symptoms within-session; and falls incidence weekly for 6 months following intervention completion. Hypothesis: At primary endpoint, participants in the experimental group will show more improvement than participants in the control group in measures sensitive to neuropathy disease state (i.e., sway variability and area).

Aim2: To evaluate change in gait variability after 16 sessions of Tango (exp) vs HEX (control) (n=26 per group; 1:1 randomization). As secondary measures, to analyze local and orbital dynamic stability (pre, post, and 1mo post-intervention), PROs (monthly), and falls incidence (weekly) following intervention completion. Hypothesis: At primary endpoint, participants in the experimental group will show more improvement than participants in the control group in measures of gait variability (i.e., stride-to-stride variability in speed).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivor stage I-III
* Symptomatic for neuropathy
* postural control outside 70% CI for adults who are middle-aged without neurotrauma
* having completed taxane-based chemotherapy treatment at least 3 months ago;
* able to understand and comply with directions associated with testing and study treatments.

Exclusion Criteria:

* Pre-existing vestibular deficit;
* poorly controlled diabetes (hgA1C > 8);
* non-ambulatory or lower extremity amputation (assistive devices allowed);
* use of cytotoxic or immunotherapy during study (endocrine therapy allowed);
* participation in physical therapy during the study;
* contraindication to participate in Tango due to orthopedic issue (e.g., herniated vertebral disc);

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Worthen-Chaudhari, PhD, MFA, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hackney ME, Earhart GM. Recommendations for Implementing Tango Classes for Persons with Parkinson Disease. Am J Dance Ther. 2010 Jun;32(1):41-52. doi: 10.1007/s10465-010-9086-y. PMID 30369677
- [Background] Zimmer P, Trebing S, Timmers-Trebing U, Schenk A, Paust R, Bloch W, Rudolph R, Streckmann F, Baumann FT. Eight-week, multimodal exercise counteracts a progress of chemotherapy-induced peripheral neuropathy and improves balance and strength in metastasized colorectal cancer patients: a randomized controlled trial. Support Care Cancer. 2018 Feb;26(2):615-624. doi: 10.1007/s00520-017-3875-5. Epub 2017 Sep 30. PMID 28963591
- [Derived] Worthen-Chaudhari L, Schnell PM, Hackney ME, Lustberg MB. Partnered dance evokes greater intrinsic motivation than home exercise as therapeutic activity for chemotherapy-induced deficits: secondary results of a randomized, controlled clinical trial. Front Psychol. 2024 Jun 19;15:1383143. doi: 10.3389/fpsyg.2024.1383143. eCollection 2024. PMID 38962217
- [Derived] Lantis K, Schnell P, Bland CR, Wilder J, Hock K, Vargo C, Glover NA, Hackney ME, Lustberg MB, Worthen-Chaudhari L. Biomechanical effect of neurologic dance training (NDT) for breast cancer survivors with chemotherapy-induced neuropathy: study protocol for a randomized controlled trial and preliminary baseline data. Trials. 2023 Sep 1;24(1):564. doi: 10.1186/s13063-023-07554-z. PMID 37658464
- [Derived] Lantis KD, Schne P, Bland CR, Wilder J, Hock K, Glover NA, Hackney ME, Lustberg MB, Worthen-Chaudhari L. Biomechanical effect of neurologic dance training (NDT) for breast cancer survivors with chemotherapy-induced neuropathy: study protocol for a randomized controlled trail and preliminary baseline data. Res Sq [Preprint]. 2023 Jun 29:rs.3.rs-2988661. doi: 10.21203/rs.3.rs-2988661/v1. PMID 37461666

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Exercise (HEX): The control group will consist of an evidence-based, structured home exercise program (HEX) based on the 8 week intervention described by Zimmer et al (2018) and recommended by physical therapists specializing in BC within our organization. This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hr training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
Period: Overall Study
Arm/Group | Tango | Home Exercise (HEX)
Started | 26 | 26
Attended Introductory Session | 23 | 22
Adhered Through 4 Weeks of Intervention | 20 | 13
Adhered Through 8 Weeks of Intervention | 17 | 10
Returned for 1 Month Follow-up Post Intervention | 17 | 8
Completed | 17 | 8
Not Completed | 9 | 18

BASELINE CHARACTERISTICS:
Groups:
- Home Exercise (HEX): The control group will consist of an evidence-based, structured home exercise program (HEX) based on the 8 week intervention described by Zimmer et al (2018) and recommended by physical therapists specializing in BC within our organization. This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hr training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
  Evidence-Based Exercise: This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hr training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
- Total: Total of all reporting groups
Arm/Group | Tango | Home Exercise (HEX) | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.37) | 58.9 (10.4) | 61.2 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Postural Control (Variability)
Description: root-mean square of the center of pressure (COP)
Time Frame: At baseline, week 8 of intervention, and at 4 week follow-up post intervention
Population: The number of participants analyzed at each time point represents the number who participated in the postural control tests at each timepoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 24
millimeters
  Baseline | 10.3 (4.93) | 9.64 (2.42)
  Week 8: number analyzed (Participants) | 18 | 10
  Week 8 | 8.03 (3.54) | 8.00 (2.82)
  Follow-up Visit (4 weeks post-intervention): number analyzed (Participants) | 18 | 11
  Follow-up Visit (4 weeks post-intervention) | 7.74 (3.67) | 8.61 (2.31)

2. Primary Outcome: Intrinsic Motivation
Description: Intrinsic motivation will be measured using a subscale of the Intrinsic Motivation Inventory (IMI). The 6 item Interest/Enjoyment subscale of the IMI represents intrinsic motivation in an activity just performed as a possible score of 6 to 36 with 6 = most; 18 = neutral; 36 = least interesting/enjoyable. Specific items queried include whether the activity just performed was: enjoyable, enjoyed, boring (reverse order), interesting, fun, and able to hold the participant's attention.
Time Frame: Assessed at week 4, week 8, and week 12
Population: The number of analyzed participants is the number of participants who were still adhering to the study intervention at the time points that intrinsic motivation data was collected
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 20 | 13
score on a scale
  4 weeks | 6 [6 to 11.5] | 21.5 [19 to 24]
  8 weeks: number analyzed (Participants) | 17 | 10
  8 weeks | 6 [6 to 8.5] | 18 [14.2 to 20]
  12 weeks: number analyzed (Participants) | 17 | 8
  12 weeks | 6 [6 to 6] | 16 [14 to 19]

3. Secondary Outcome: Postural Control (Ellipse Area)
Description: 95% ellipse area of the COP
Time Frame: At baseline, week 8 of intervention, and at 4 week follow-up post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared
Groups:
- Tango (TEX): The intervention will consist of 16 Argentine Tango (Tango) sessions, adapted for neurorehabilitation per Hackney and Earhart (2010). Delivered over 8 weeks at a frequency of 2x per week and duration of 1 hour per session, this program teaches the basics steps of partnered Tango dance.
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 24
millimeters squared
  Baseline | 1023 (1052) | 775 (441)
  Week 8: number analyzed (Participants) | 25 | 10
  Week 8 | 595 (618) | 574 (389)
  Follow-up Visit (4 weeks post-intervention): number analyzed (Participants) | 25 | 11
  Follow-up Visit (4 weeks post-intervention) | 570 (606) | 647 (323)

4. Secondary Outcome: Postural Control (Velocity)
Description: velocity of COP
Time Frame: At baseline, week 8 of intervention, and at 4 week follow-up post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters per second
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 24
millimeters per second
  Baseline | 10.2 (6.31) | 12.1 (5.86)
  Week 8: number analyzed (Participants) | 18 | 10
  Week 8 | 7.51 (3.56) | 7.92 (4.12)
  Follow-up Visit (4 weeks post-intervention): number analyzed (Participants) | 18 | 11
  Follow-up Visit (4 weeks post-intervention) | 9.21 (5.99) | 8.64 (2.79)

5. Secondary Outcome: Postural Control (Complexity)
Description: sample entropy of the center of pressure (COP). Sample entropy is a non-linear COP measure that determines the irregularity of a time-series. Sample entropy of the resultant COP position will be calculated using the increment calculation method (SEI) with constant values applied of m = 3 and r = 0.3. Entropy of postural responses represents the automatic complexity of neuromotor control that is available to an individual. Sample entropy scores won't go below 0 or above 2, and higher values indicate better complexity in postural response
Time Frame: At baseline, week 8 of intervention, and at 4 week follow-up post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sample entropy score
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 24
sample entropy score
  Baseline | 0.480 (0.157) | 0.467 (0.120)
  Week 8: number analyzed (Participants) | 18 | 10
  Week 8 | 0.558 (0.161) | 0.566 (0.124)
  Follow-up Visit (4 weeks post-intervention): number analyzed (Participants) | 18 | 11
  Follow-up Visit (4 weeks post-intervention) | 0.559 (0.121) | 0.559 (0.103)

6. Secondary Outcome: Postural Control (Variability) at Tango Sessions
Description: root-mean square of the center of pressure (COP). The mean will be taken of all beginning of session data points together and all end of session data points together. Lower numbers indicate better neuromotor health.
Time Frame: at the beginning and at the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: Postural control at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 0
millimeters
  Beginning of Sessions | 8.86 (4.43) |
  End of Sessions | 8.74 (4.48) |

7. Secondary Outcome: Postural Control (Ellipse Area) at Tango Sessions
Description: 95% ellipse area of the COP. The mean will be taken of all beginning of session data points together and all end of session data points together. Lower numbers indicate better neuromotor health.
Time Frame: at the beginning and at the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: Postural control at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 0
millimeters squared
  Beginning of Sessions | 749 (874) |
  End of Sessions | 748 (856) |

8. Secondary Outcome: Postural Control (Velocity) at Tango Sessions
Description: velocity of COP. The mean will be taken of all beginning of session data points together and all end of session data points together. Lower numbers indicate better neuromotor health.
Time Frame: at the beginning and the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: Postural control at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: millimeters per second
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 0
millimeters per second
  Beginning of Sessions | 8.87 (5.33) |
  End of Sessions | 8.08 (4.37) |

9. Secondary Outcome: Postural Control (Complexity) at Tango Sessions
Description: sample entropy of the center of pressure (COP). Sample entropy is a non-linear COP measure that determines the irregularity of a time-series. Sample entropy of the resultant COP position will be calculated using the increment calculation method (SEI) with constant values applied of m = 3 and r = 0.3. Entropy of postural responses represents the automatic complexity of neuromotor control that is available to an individual. Sample entropy scores won't go below 0 or above 2, and higher values indicate better complexity in postural responseThe mean will be taken of all beginning of session data points together and all end of session data points together
Time Frame: at the beginning and the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: Postural control at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: sample entropy score
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 25 | 0
sample entropy score
  Beginning of Sessions | 0.520 (0.145) |
  End of Sessions | 0.546 (0.180) |

10. Secondary Outcome: Clinical Measure of Balance Function
Description: The Timed Up-and-Go test, or TUG, (<2 min to administer) is a timed test of a person's ability to stand from a chair, walk 10 feet, turn around, and return to sitting with shorter times indicating better functional balance.
Time Frame: At baseline, week 4 of intervention, and at 4 week follow-up post intervention, up to 12 weeks
Population: The number of participants analyzed represents the number who completed the TUG tests at each timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 16 | 10
seconds
  Baseline: number analyzed (Participants) | 5 | 7
  Baseline | 10.3 (2.47) | 11.7 (5.21)
  Week 4: number analyzed (Participants) | 14 | 8
  Week 4 | 8.65 (1.92) | 8.25 (1.74)
  Follow-up Visit (4 weeks post-intervention) | 8.49 (1.79) | 7.70 (1.25)

11. Secondary Outcome: Neuropathy Symptoms Score at Tango Sessions
Description: European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire, Chemotherapy-Induced Peripheral Neuropathy (CIPN 20): is a validated instrument for longitudinal evaluation of neuropathy symptoms induced by chemotherapy. This is a 20-item patient reported questionnaire. It is easy to use and filled out by patients themselves. Scores range between 1 to 10 with higher scores indicating greater chemotherapy-induced peripheral neuropathy (CIPN) severity. The mean will be taken of all beginning of session data points together and all end of session data points together
Time Frame: at the beginning and the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: Neuropathy symptoms scores at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 22 | 0
score on a scale
  Beginning of sessions | 6.68 (4.25) |
  End of sessions | 3.29 (3.01) |

12. Secondary Outcome: Neuropathy Symptoms Score
Description: European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire, Chemotherapy-Induced Peripheral Neuropathy (CIPN 20): is a validated instrument for longitudinal evaluation of neuropathy symptoms induced by chemotherapy. This is a 20-item patient reported questionnaire. It is easy to use and filled out by patients themselves. Scores range between 1 to 10 with higher scores indicating greater chemotherapy-induced peripheral neuropathy (CIPN) severity.
Time Frame: At week 8 of intervention and at 4-week follow-up post intervention
Population: The number of participants analyzed is the number of participants for which neuropathy symptoms scores were collected at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 20 | 10
score on a scale
  Week 8 | 6.60 (3.97) | 6.89 (7.41)
  Follow-up (4 weeks post-intervention): number analyzed (Participants) | 18 | 10
  Follow-up (4 weeks post-intervention) | 7.06 (4.08) | 5.18 (5.36)

13. Secondary Outcome: Brief Pain Inventory Short Form at Tango Sessions
Description: The Brief Pain Inventory Short Form (BPI) is a validated instrument used to evaluate pain symptoms and functional capacity "right now" using a single item visual analog scale (VAS) on which participants will rate how much pain they are in "right now" on a scale of 1 to 10 (10 being high the worst pain imaginable). The mean will be taken of all beginning of session data points together and all end of session data points together
Time Frame: at the beginning and the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: BPI scores at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 23 | 0
score on a scale
  Beginning of sessions | 1.68 (1.59) |
  End of sessions | 1.20 (1.28) |

14. Secondary Outcome: Brief Pain Inventory Short Form
Description: The Brief Pain Inventory Short Form (BPI) is a validated instrument used to evaluate pain symptoms and functional capacity "right now" using a single item visual analog scale (VAS) on which participants will rate how much pain they are in "right now" on a scale of 1 to 10 (10 being high the worst pain imaginable).
Time Frame: At week 8 of intervention and at 4-week follow-up post intervention
Population: The number of participants analyzed is the number of participants for which BPI scores were collected at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 20 | 10
score on a scale
  Week 8 | 1.72 (1.53) | 1.07 (0.999)
  Follow-up (4 weeks post-intervention): number analyzed (Participants) | 18 | 10
  Follow-up (4 weeks post-intervention) | 1.78 (1.83) | 1.55 (1.99)

15. Secondary Outcome: Cancer-Related Fatigue (BFI Scores) at Tango Sessions
Description: The Brief Fatigue Inventory (BFI) is used to rapidly assess the severity and impact of cancer-related fatigue "right now" using a single item visual analog scale (VAS) on which participants will rate how much fatigue they feel "right now" on a scale of 1 to 10 (10 being high the worst fatigue imaginable). The mean will be taken of all beginning of session data points together and all end of session data points together
Time Frame: at the beginning and the end of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Population: BFI scores at Tango sessions were only measured for participants in the Tango arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 23 | 0
score on a scale
  Beginning of sessions | 8.56 (9.61) |
  End of sessions | 1.21 (1.30) |

16. Secondary Outcome: Cancer-Related Fatigue
Description: The Brief Fatigue Inventory (BFI) is used to rapidly assess the severity and impact of cancer-related fatigue "right now" using a single item visual analog scale (VAS) on which participants will rate how much fatigue they feel "right now" on a scale of 1 to 10 (10 being high the worst fatigue imaginable).
Time Frame: At week 8 and at 4-week follow-up visit post intervention
Population: The number of participants analyzed is the number of participants for which BFI scores were collected at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tango (TEX) | Home Exercise (HEX)
Number analyzed (Participants) | 20 | 10
score on a scale
  Week 8 | 8.13 (8.95) | 10.7 (11.4)
  Follow-up (4 weeks post intervention): number analyzed (Participants) | 18 | 9
  Follow-up (4 weeks post intervention) | 7.22 (8.72) | 13.3 (14.3)

17. Secondary Outcome: Number of Falls
Description: the number of falls or near falls that the participant remembers experiencing in the month prior to enrollment in the study will be assessed. All reported falls will be totaled and reported by arm.
Time Frame: once at the point of study enrollment
Measure: Number; unit: number of falls
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 26 | 26
number of falls | 1 | 0

18. Secondary Outcome: Number of Falls
Description: the number of falls or near falls experienced by the participant since last evaluation/intervention session. All reported falls throughout the intervention time period will be totaled and reported by arm.
Time Frame: at the beginning of each assessment or intervention session for up to 20 sessions, up to 8 weeks
Measure: Number; unit: Number of falls
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 26 | 26
Number of falls | 1 | 0

19. Secondary Outcome: Number of Falls
Description: the number of falls or near falls experienced by the participant in the 6 months post-intervention. All reported falls throughout the follow-up time period will be totaled and reported by arm
Time Frame: 6 months post-intervention
Measure: Number; unit: Number of falls
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 26 | 26
Number of falls | 0 | 1

20. Secondary Outcome: Change in Dual-task Function
Description: Dual task function was measured using the Timed-Up-and-Go motor task while counting backward by 3 s (TUGCog), a validated clinical test of dual-task function for which lower values indicate better performance. To perform this test, participants completed the Timed-Up-and Go (TUG) test commonly used in clinical practice wherein individuals stand from a chair with arms, walk 3 meters, turn around, and return to sitting as fast as safely possible (i.e. motor task) while counting out loud and backward by 3 s (i.e. cognitive task). The test is completed 3 times, with rest allowed between trials. Time in seconds per trial is averaged to produce the TUGCog score per timepoint.
Time Frame: Assessed at baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Home Exercise (HEX): The control group will consist of an evidence-based, structured home exercise program (HEX) based on the 8 week intervention described by Zimmer et al (2018) and recommended by physical therapists specializing in BC within our organization. This program consists of information on neuropathy and fall prevention combined with a schedule of 1 hour training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
  Evidence-Based Exercise: This program consists of information on neuropathy and fall prevention combined with a schedule of 45 minute training (i.e., endurance, resistance, and sensorimotor) performed 2x per week
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 26 | 26
seconds
  Change between baseline to 4 weeks | -2.65 [-3.37 to -1.94] | -1.9 [-2.77 to -1.03]
  Change between baseline and 8 weeks | -2.47 [-3.16 to -1.78] | -2.65 [-3.52 to -1.77]
  Change between baseline and 12 weeks (follow-up visit) | -2.68 [-3.51 to -1.84] | -3.06 [-3.96 to -2.16]

21. Secondary Outcome: Adherence
Description: Adherence is measured by the number of enrollees who participated through each time point of the study
Time Frame: Assessed at baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Number; unit: participants
Arm/Group | Tango | Home Exercise (HEX)
Number analyzed (Participants) | 26 | 26
participants
  Randomized | 26 | 26
  Attended Introductory Session | 23 | 22
  Adhered through 4 weeks of intervention | 20 | 13
  Adhered through 8 weeks of intervention | 17 | 10
  Returned for follow-up 1 month post- intervention (12 week timepoint) | 17 | 8

22. Other Pre Specified Outcome: Quantified Clinical Measure of Balance Function
Description: The Mini Balance Evaluation System Test short version (MiniBEST): evaluates sensory organization, anticipatory and reactive postural control, and dynamic gait indices on a scale from 1 to 28 points (28 represents the highest function measurable by the test); was recently recommended for use in studies of neuropathy; and discriminated BC survivors from controls in at least 1 prior study. Instrumentation of MiniBEST will enable the calculation of spatiotemporal, kinematic, and co-contraction measures
Time Frame: 8 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Quantified Clinical Measure of Balance Function
Description: as for outcome 22
Time Frame: 1 month follow-up post-intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Tango (TEX) | Home Exercise (HEX)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/26
Other Adverse Events (participants affected / at risk) | 19/26 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tango (TEX) (N=26) | Home Exercise (HEX) (N=26)
Hospitalized due to low hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalized due to fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalized due to fall with broken wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tango (TEX) (N=26) | Home Exercise (HEX) (N=26)
Ankle pain (possibly tendonitis per Dr) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID+ (Infections and infestations) | 3 (3) | 2 (2)
Fall/LOB- uninjured (Injury, poisoning and procedural complications) | 6 (27) | 2 (2)
Feeling unwell/ cold (General disorders) | 4 (6) | 7 (10)
GI distress (Gastrointestinal disorders) | 1 (1) | 1 (2)
Head cold sinuses (Infections and infestations) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection Axilla (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection Sinus/Ear (Infections and infestations) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Planned surgery: chemo port removed (Surgical and medical procedures) | 1 (1) | 0 (0)
Planned surgery: melanoma removed (Surgical and medical procedures) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Poison ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shoulder pain during tango INT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 1 (1)
Stress fracture hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thumb strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tripped; would have fallen if son-in-law hadn't caught (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccine reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Walking pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Broken toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Endoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Knee arthritis pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left hip discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Long COVID headache (Nervous system disorders) | 0 (0) | 1 (1)
Nerve pain (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinus infection and symptoms of POTS (Infections and infestations) | 0 (0) | 1 (1)
Steroid injection for foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Symptoms of Postural Orthostatic Tachycardia Syndrome (POTS) (Cardiac disorders) | 0 (0) | 1 (1)
Trauma to toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT05114005/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT05114005/ICF_001.pdf